CLINICAL TRIAL: NCT04810832
Title: EXPRESON-INTRA : Intracerebral Recordings of P3a Responses to Own-names Uttered by Expressive and Neutral Voices in Pharmacoresistant Epilepsy Adult Patients
Brief Title: EXPRESON-IN : Intracerebral Recordings of P3a Responses to Expressive Own-names
Acronym: EXPRESON-IN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A01340-39
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-01

CONDITIONS: Intractable Epilepsy
Keywords: Event-related Potentials (ERP); Intracerebral recordings; Presurgical evaluation
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: Open and prospective study.
  Evoked related potentials are recorded on the scalp and with intracranial electrodes for each participant while they listen 3 paradigms successively and in a random order:
  i) their own name uttered by a smiling voice ii) their own name uttered by a neutral voice iii) their own name uttered by a rough voice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole group (Experimental): The whole group undergo the two phases of the study:
  * 1/ They listen successively the 3 oddball paradigms in the department of neurophysiology : P3 own-name recorded by listening to a smiling voice P3 own-name recorded by listening to a neutral voice P3 own-name recorded by listening to a rough voice
  * 2/ They listen successively the same 3 oddball paradigms in the neurosurgical department, during their intractable epilepsy presurgical evaluation : P3 own-name recorded by listening to a smiling voice P3 own-name recorded by listening to a neutral voice P3 own-name recorded by listening to a rough voice
  Interventions: Other: Evoked related potentials

INTERVENTIONS:
Other: Evoked related potentials — Evoked related potentials are performed for each patient during each paradigm (neutral voice and expressive voices):
  * with scalp electrodes in the department of neurophysiology
  * with intracranial electrodes in the department of neurosurgery.

SUMMARY:
Neurophysiologic evaluation of disorders of consciousness (DOC) patients in intensive care unit include late auditory evoked potentials. It allows the physicians to record cerebral responses of patients to auditory stimuli and in particularly to their own name (as the P3a response). Numerous studies try to improve the relevance of the auditory stimuli used in this paradigm and notably using more expressive stimuli.

Here the investigators investigate the intracerebral correlates of the P3a responses recorded on the scalp with neutral and more expressive stimuli.

DETAILED DESCRIPTION:
Late auditory evoked potentials (as P3 wave) are used in neurophysiology to assess the level of consciousness in DOC (disorder of consciousness) patients. The P3 wave, elicited by listening standard and deviant stimuli, corresponds to the activation of a frontoparietal network and is considered to reflect a cognitive attention task. Using the own name of the patient as deviant stimuli improve the ability to detect the P3 wave because of the particularly relevance of this stimulus for the patient.

In human cognition, to identify the expressivity valence of a voice is essential. Neural processing of expressive voices should involves more widespread brain areas than neutral voices processing.

Here the investigators investigate the intracerebral correlates of the P3a responses recorded on the scalp to own-name stimuli uttered by neutral and more expressive voices (positive : smiling voice or negative : rough voice) in adult pharmacoresistant epilepsy patients.

ELIGIBILITY:
Inclusion Criteria:

* Intractable focal epilepsy with undergoing pre-surgical evaluation
* intracerebral electrodes implantation in auditory cortices, temporal lobe, superior temporal gyrus, limbic areas, frontal lobe
* Given Consent to inclusion

Exclusion Criteria:

* Deafness
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-09-09 (Estimated); Study Completion 2023-09-09 (Estimated)

PRIMARY OUTCOMES:
Latencies cartography of intracranial responses to own-name uttered by neutral voice | 1 year
  Analyse of latencies of intracranial responses recorded to own-name uttered by neutral voice to build a map of the brain process of this responses
Latencies cartography of intracranial responses to own-name uttered by expressive voices | 1 year
  Analyse of latencies of intracranial responses recorded to own-name uttered by expressive voices to build a map of the brain process of this responses

SECONDARY OUTCOMES:
Comparison between brain responses to own-name uttered by expressive voices recorded with intracerebral electrodes versus scalp electrodes | 1 year
  Qualitative comparison between scalp and intracranial recordings with the expressive voices paradigms (comparison of the latencies of the recorded responses)
Comparison between brain responses to own-name uttered by neutral voices recorded with intracerebral electrodes versus scalp electrodes | 1 year
  Qualitative comparison between scalp and intracranial recordings with the neutral voices paradigms (comparison of the latencies of the recorded responses)

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Paris - Sainte Anne, Paris, France